CLINICAL TRIAL: NCT03465605
Title: Frailty Assesment in the Congestive Heart Failure Clinic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0072-17MMC
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Fragility Syndrome; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: frailty test — questionnaire

SUMMARY:
Frailty is known as an independent risk factor for morbidity and mortality in older cardiac patients, including patients with congestive heart failure. It is an important factor taken into the cardiologists decision making in the clinic, and influences the intensity of follow up treatment, invasive intervention and the need to ensure a stronger social support system for the patient. Frailty assessment is usually made subjectively by the cardiologist, known in the literature as eyeball testing.

In this study the investigators will compare the cardiologists subjective eyeball testing to objective frailty assessment tests based on Fried score and Edmonton frail scale

DETAILED DESCRIPTION:
Elderly patients visiting the congestive heart failure clinic at Meir Medical Center will be assessed for frailty twice. Once in an "eyeball" test by their cardiologist at the clinic, and a second time in an objective test based on fried and Edmonton frailty scores.

The second subjective assessment will be made by geriatric and internal medicine physicians, and the cardiologist won't be aware of the results of the objective assessment.

The results of both tests will be compared.

ELIGIBILITY:
Inclusion Criteria:

* patients an the Meir congestive heart failure clinic.
* age 70 and above
* can sign an informed consent

Exclusion Criteria:

* patients admitted in the last two month

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 70 years old and older visiting the congestive heart failure clinic at the Meir Medical Center, who can sign an informed consent and hasn't been admitted to the hospital in the past two month.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
An objective frailty assessment using fries score an Edmonton frailty scale will be compared to a subjective eyeball frailty assessment. | 1 week

IPD SHARING:
Plan to Share IPD: Yes